CLINICAL TRIAL: NCT03505359
Title: Post-operative Rehabilitation Protocol for Combined Reconstruction of Anterior Cruciate Ligament and Anterolateral Knee Ligament Surgery
Brief Title: Rehabilitation Protocol for Reconstruction of Anterior Cruciate Ligament and Anterolateral Knee Ligament Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Silvia Maria Amado João, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54541116.8.0000.0068
Record Dates: First submitted 2017-10-03; First posted 2018-04-23 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Anterolateral Ligament Reconstruction; Rehabilitation

STUDY DESIGN:
Intervention Model Description: A blinded randomized clinical trial will be conducted to evaluate the effects of two protocols for the rehabilitation of patients undergoing combined re-construction of ACL and ALL.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Group treated by the new protocol with partial knee immobilization
  Interventions: Other: partial knee immobilization protocol
- Control group (Active Comparator): Group treated by a standard protocol for ACL reconstruction.
  Interventions: Other: standard ACL reconstruction rehabilitation protocol

INTERVENTIONS:
Other: partial knee immobilization protocol — 12 weeks rehabilitation protocol including exercises to improve range of motion, gait, balance, muscle strength with a 0-60 degrees articulated knee brace in the first 6 weeks in the experimental group.
  Arms: Experimental group
Other: standard ACL reconstruction rehabilitation protocol — 12 weeks rehabilitation protocol including exercises to improve range of motion, gait, balance, muscle strength.
  Arms: Control group

SUMMARY:
Introduction: Individuals with an ACL lesion present abnormal rotational stability. Among the structures located in the anterolateral region of the knee that could act as restraints of the rotational knee lassitude, there is the Anterior Lateral Ligament (ALL), and its reconstruction associated with ACL reconstruction could reduce recurrence injury rates. Objective: to develop a rehabilitation protocol for patients undergoing combined reconstruction of ACL and ALL. METHOD: Articles published with patients submitted to ACL reconstruction with an anatomic technique and flexor tendon graft, (which is the same one adopted in this study), were selected as a base to this protocol. Discussion: The results will provide important information on clinical practice, since it can help identify the necessity or not of restraining the knee range of motion in combined surgeries. It can guide the therapeutic planning, including the cost of knee restraint devices, in addition to estimating these patients prognosis. The protocol with partial restriction of knee range of motion in the first 6 weeks of postoperative is the most indicated program in the rehabilitation of the combined surgeries of ACL and ALL reconstruction.

DETAILED DESCRIPTION:
Currently, the anatomical reconstruction of the ACL has been widely used, with the purpose of increasing the knee rotational control after the injury, and thus, to improve the clinical evolution in the long term. The concept involves restoring knee kinematics by improving function by reducing the number of graft failures, delaying or preventing degeneration of the joint. Normally, rehabilitation protocols in these cases are more careful with respect to knee ROM gain and use of exercises in open kinetic chain, with the purpose of preserving the graft.

Allied to this concept, the use of extra-articular reconstruction associated with ACL reconstruction, gained new horizons with the discovery of ALL, signaling to the possibility of a better rotational control and, consequently, a decrease in the number of graft failures.

Due to the particularities of each surgical technique, it is necessary that the rehabilitation protocols adapt to the different methods, guaranteeing the functional recovery, but without damages to the reconstruction.

With the proposal of ACL reconstruction surgery associated with ALL reconstruction, it is necessary to develop a specific rehabilitation protocol for these patients, considering some postoperative specificities of extra-articular reconstructions, since they are data that are not available in the literature until now.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged from 18 to 40 years
* Documented and symptomatic anterior cruciate ligament (ACL) injury followed by ACL+ anterolateral ligament (ALL) ligament reconstruction

Exclusion Criteria:

* Patients with multiple ligament injuries
* Bilateral ACL injury

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male individuals will be selected to avoid physiological differences between genders, such as muscle strength, flexibility and ligamentous laxity.
Enrollment: 28 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
Knee Function | 12 months
  Lysholm Knee Scoring Scale: instrument consisting of eight domains: limping, support, re-straining, instability, pain, swelling, climbing stairs and squatting, with closed-answers alternatives. The final result is expressed in nominal and ordinal form, being "excellent" ranging from 95 to 100 points; "Good" from 84 to 94 points; "Regular" between 65 and 83 and "bad" when values are equal to or less than 64.

SECONDARY OUTCOMES:
Follow-up of knee function | 3 weeks; 6 weeks; 12 weeks; 6 months
  Lysholm Knee Scoring Scale: instrument consisting of eight domains: limping, support, re-straining, instability, pain, swelling, climbing stairs and squatting, with closed-answers alternatives. The final result is expressed in nominal and ordinal form, being "excellent" ranging from 95 to 100 points; "Good" from 84 to 94 points; "Regular" between 65 and 83 and "bad" when values are equal to or less than 64.
Static Postural Control | 3 weeks; 6 weeks; 12 weeks; 6 months and 12 months
  Static Postural Control will be assessed through the AccuSuway mobile power platform.(AMTI®).
Dynamic Postural Control | 3 weeks; 6 weeks; 12 weeks; 6 months and 12 months
  Dynamic Postural Control will be assessed through the Balance Master System (BMS) platform.
Muscle strength | 3 weeks; 6 weeks; 12 weeks; 6 months and 12 months
  The isometric and isokinetic strength test will be performed by an isokinetic dynamometry (Biodex Multi-Joint System III), used to record the torque of the knee flexor and extensor muscles, as well as the hip abductors.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia M João, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- USaoPauloGH, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available until the protocol is published